CLINICAL TRIAL: NCT04378712
Title: Effects of Hydrogen/Oxygen Mixed Gas Inhalation for Patients With Coronavirus Disease 2019 (COVID-19) Who Had Dyspnea: A Multicenter, Open-label Clinical Trial
Brief Title: Hydrogen/Oxygen Mixed Gas Inhalation for Coronavirus Disease 2019 (COVID-19)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Responsible Party: Principal Investigator, Weijie Guan, Associate professor of respiratory medicine, co-principal investigator, Guangzhou Institute of Respiratory Disease
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JT202005LZ
Record Dates: First submitted 2020-04-29; First posted 2020-05-07 (Actual); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: Covid-19; Hydrogen/Oxygen Mixed Gas; Dyspnea
Keywords: Covid-19; Hydrogen/oxygen mixed gas; Dyspnea
MeSH Terms: conditions — COVID-19; Dyspnea | interventions — Nebulizers and Vaporizers; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): H2-O2 (66% hydrogen; 33% oxygen) inhalation. Patients in treatment group inhaled H2-O2 (66% hydrogen; 33% oxygen) at 3 L/min via nasal cannula by using the Hydrogen/Oxygen Generator (model AMS-H-03, Shanghai Asclepius Meditech Co., Ltd., China) until discharge.
  Interventions: Device: Hydrogen Oxygen Generator with Nebulizer; Other: Standard-of-care
- Control Group (Other): Usual care referred to the standard-of-care (including oxygen therapy) recommended by Chinese National Health Commission.
  Interventions: Other: Standard-of-care

INTERVENTIONS:
Device: Hydrogen Oxygen Generator with Nebulizer — Patients in treatment group inhaled H2-O2 (66% hydrogen; 33% oxygen) at 3 L/min via nasal cannula by using the Hydrogen/Oxygen Generator (model AMS-H-03, Shanghai Asclepius Meditech Co., Ltd., China) until discharge.
  Arms: Intervention Group
Other: Standard-of-care — Standard-of-care consisted of the supportive therapies (including oxygen therapy) recommended by the Chinese National Health Commission

SUMMARY:
This was a randomized, multi-center, open-label clinical trial. Eligible patients were recruited from seven hospitals in China. On the basis of standard-of-care, patients in treatment group inhaled H2-O2 (66% hydrogen; 33% oxygen) at 3 L/min via nasal cannula by using the Hydrogen/Oxygen Generator (model AMS-H-03, Shanghai Asclepius Meditech Co., Ltd., China) until discharge. Patients in control group received standard-of-care (consisting of oxygen therapy) alone until discharge.

DETAILED DESCRIPTION:
This was a randomized, multi-center, open-label clinical trial. Eligible patients were recruited from seven hospitals in China. On the basis of standard-of-care, patients in treatment group inhaled H2-O2 (66% hydrogen; 33% oxygen) at 3 L/min via nasal cannula by using the Hydrogen/Oxygen Generator (model AMS-H-03, Shanghai Asclepius Meditech Co., Ltd., China) until discharge. Patients in control group received standard-of-care (consisting of oxygen therapy) alone until discharge. Clinical assessments included the five-category ordinal scale, four-category ordinary scale of dyspnea, coughing, chest distress and chest pain (0: None; 1: Mild; 2: Moderate; 3: Severe; 4: Very severe) and adverse events, performed on admission, at enrollment, at day 2 and 3 after randomization, and the day before discharge. The primary endpoint was the proportion of patients with improved disease severity (by at least one scale). Secondary endpoints comprised the change from baseline in oxygen saturation and symptom scales.

ELIGIBILITY:
Inclusion Criteria:

* Patients with lab-confirmed Covid-19 aged 18 to 75 years.
* Had dyspnea both on hospital admission and at enrollment.
* The patients volunteered to participate in this study and signed the informed consent

Exclusion Criteria:

* Have other systemic diseases other than COVID-19 -- a disease that, according to the investigator's judgment, might increase the risk of developing adverse outcomes or affect the outcome measures after participation in the study.

Women who are pregnant or breastfeeding or plan to be pregnant during the study.

Subjects with one of the following respiratory diseases:

* Subjects in critical or unstable conditions. Critical (meeting any of the following symptoms): 1. Respiratory failure occurs and mechanical ventilation is needed; 2. Shock occurs; 3. Other organ failure, ICU monitoring and treatment is needed.
* Having immunosuppressive diseases (HIV), severe neurological disease affecting upper respiratory tract control, or other risk factors that the investigator believes can cause a significant risk of pneumonia in subjects.
* Subjects with mental disorder and cognitive impairment.
* Subjects who do not follow the study steps.
* Patients with mental retardation, poor motivation, drug abuse (including drugs and alcohol) or other disease history restricting the effectiveness of informed consent in this study.
* Use of antioxidants, including large doses of vitamin C and vitamin E.
* Subjects who are not suitable for participation in this study in the judgment of investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2020-01-21 (Actual); Primary Completion 2020-03-23 (Actual); Study Completion 2020-03-23 (Actual)

PRIMARY OUTCOMES:
The proportion of patients with improved disease severity at day 2 | from baseline to day 2
  The proportion of patients with improved disease severity (by at least one scale) at day 2
The proportion of patients with improved disease severity at day 3 | from baseline to day 3
  The proportion of patients with improved disease severity (by at least one scale) at day 3
The proportion of patients with improved disease severity at the day before hospital discharge | up to 14 days (from baseline to the day before hospital discharge)
  The proportion of patients with improved disease severity (by at least one scale) at the day before hospital discharge

SECONDARY OUTCOMES:
The change from baseline in oxygen saturation at day 2. | from baseline to day 2
  The change from baseline in oxygen saturation at day 2.
The change from baseline in oxygen saturation at day 3. | from baseline to day 3
  The change from baseline in oxygen saturation at day 3.
The change from baseline in oxygen saturation at the day before hospital discharge | up to 14 days (from baseline to the day before hospital discharge)
  The change from baseline in oxygen saturation at the day before hospital discharge.
The change from baseline in dyspnea scale at day 2. | from baseline to day 2
  The change from baseline in dyspnea scale (ranging from 0-4, with higher scores indicating severer outcomes) at day 2.
The change from baseline in dyspnea scale at day 3. | from baseline to day 3
  The change from baseline in dyspnea scale (ranging from 0-4, with higher scores indicating severer outcomes) at day 3.
The change from baseline in dyspnea scale at the day before hospital discharge. | up to 14 days (from baseline to the day before hospital discharge)
  The change from baseline in dyspnea scale (ranging from 0-4, with higher scores indicating severer outcomes) at the day before hospital discharge.
The change from baseline in cough scale at day 2 | from baseline to day 2
  The change from baseline in cough scale (ranging from 0-4, with higher scores indicating severer outcomes) at day 2
The change from baseline in cough scale at day 3 | from baseline to day 3
  The change from baseline in cough scale (ranging from 0-4, with higher scores indicating severer outcomes) at day 3
The change from baseline in cough scale at the day before hospital discharge | up to 14 days (from baseline to the day before hospital discharge)
  The change from baseline in cough scale (ranging from 0-4, with higher scores indicating severer outcomes) at the day before hospital discharge
The change from baseline in chest pain scale at day 2. | from baseline to day 2
  The change from baseline in chest pain scale (ranging from 0-4, with higher scores indicating severer outcomes) at day 2.
The change from baseline in chest pain scale at day 3. | from baseline to day 3
  The change from baseline in chest pain scale (ranging from 0-4, with higher scores indicating severer outcomes) at day 3.
The change from baseline in chest pain scale at the day before hospital discharge. | up to 14 days (from baseline to the day before hospital discharge)
  The change from baseline in chest pain scale (ranging from 0-4, with higher scores indicating severer outcomes) at the day before hospital discharge.
The change from baseline in chest distress scale at day 2. | from baseline to day 2
  The change from baseline in chest distress scale (ranging from 0-4, with higher scores indicating severer outcomes) at day 2.
The change from baseline in chest distress scale at day 3. | from baseline to day 3
  The change from baseline in chest distress scale (ranging from 0-4, with higher scores indicating severer outcomes) at day 3.
The change from baseline in chest distress scale at the day before hospital discharge. | up to 14 days (from baseline to the day before hospital discharge)
  The change from baseline in chest distress scale (ranging from 0-4, with higher scores indicating severer outcomes) at the day before hospital discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Wei-jie Guan, PhD, Principal Investigator — Guangzhou Institute of Respiratory Disease
Locations (1):
- First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wu C, Chen X, Cai Y, Xia J, Zhou X, Xu S, Huang H, Zhang L, Zhou X, Du C, Zhang Y, Song J, Wang S, Chao Y, Yang Z, Xu J, Zhou X, Chen D, Xiong W, Xu L, Zhou F, Jiang J, Bai C, Zheng J, Song Y. Risk Factors Associated With Acute Respiratory Distress Syndrome and Death in Patients With Coronavirus Disease 2019 Pneumonia in Wuhan, China. JAMA Intern Med. 2020 Jul 1;180(7):934-943. doi: 10.1001/jamainternmed.2020.0994. PMID 32167524
- [Background] Xu Z, Shi L, Wang Y, Zhang J, Huang L, Zhang C, Liu S, Zhao P, Liu H, Zhu L, Tai Y, Bai C, Gao T, Song J, Xia P, Dong J, Zhao J, Wang FS. Pathological findings of COVID-19 associated with acute respiratory distress syndrome. Lancet Respir Med. 2020 Apr;8(4):420-422. doi: 10.1016/S2213-2600(20)30076-X. Epub 2020 Feb 18. No abstract available. PMID 32085846
- [Background] Zhou ZQ, Zhong CH, Su ZQ, Li XY, Chen Y, Chen XB, Tang CL, Zhou LQ, Li SY. Breathing Hydrogen-Oxygen Mixture Decreases Inspiratory Effort in Patients with Tracheal Stenosis. Respiration. 2019;97(1):42-51. doi: 10.1159/000492031. Epub 2018 Sep 18. PMID 30227423
- [Background] Morgan SE, Vukin K, Mosakowski S, Solano P, Stanton L, Lester L, Lavani R, Hall JB, Tung A. Use of heliox delivered via high-flow nasal cannula to treat an infant with coronavirus-related respiratory infection and severe acute air-flow obstruction. Respir Care. 2014 Nov;59(11):e166-70. doi: 10.4187/respcare.02728. Epub 2014 Aug 12. PMID 25118308
- [Background] Kneyber MC, van Heerde M, Markhorst DG, Plotz FB. Mechanical ventilation with heliox decreases respiratory system resistance and facilitates CO2 removal in obstructive airway disease. Intensive Care Med. 2006 Oct;32(10):1676-7. doi: 10.1007/s00134-006-0348-6. Epub 2006 Aug 23. No abstract available. PMID 16927073